CLINICAL TRIAL: NCT00681811
Title: A Multi-center, Open-Label Extension Study of HGT-1111 (Recombinant Human Arylsulfatase A or rhASA) Treatment in Patients With Late Infantile Metachromatic Leukodystrophy (MLD)
Brief Title: Open-Label Extension Study of Recombinant Human Arylsulfatase A (HGT-1111) in Late Infantile MLD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated prior to planned completion date due to lack of efficacy.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGT-MLD-049; 2008-000084-41 (EudraCT Number)
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Results first posted 2013-11-08 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Late Infantile Metachromatic Leukodystrophy
Keywords: Metazyme; Late Infantile Metachromatic Leukodystrophy
MeSH Terms: conditions — Leukodystrophy, Metachromatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HGT-1111 100 U/kg (Experimental)
  Interventions: Drug: HGT-1111
- HGT-1111 200 U/kg (Experimental)
  Interventions: Drug: HGT-1111

INTERVENTIONS:
Drug: HGT-1111 — Patients currently dosed with 100 U/kg or 200 U/kg will continue this treatment. Patients dosed with 50 U/kg will be equally randomized to treatment on 100 U/kg or 200 U/kg. The dose will be adjusted every 6-week to account for changes in body weight.The infusion length will be dependent on the dose. Infusion of 100 U/kg will be diluted in 50 ml isotonic sodium chloride and infused over 30 minutes. Infusion of 200 U/kg will be administered in the same manner except for an infusion time of 60 minutes.
  Other Names: rhASA, Metazym

SUMMARY:
This is a multi-center, open-label, extension study of patients with late infantile MLD who have previously completed clinical study HGT-MLD-048 (NCT00633139), defined as the completion of all Week 52 procedures. This group of patients will be offered ongoing treatment with HGT-1111 in this protocol. One infusion will be given every other week until the product is commercially available, the patient discontinues, or the study is terminated by the Sponsor, provided no safety issues have emerged.

DETAILED DESCRIPTION:
The primary objective of this study is to provide ongoing treatment of HGT-1111 to patients who have completed study HGT-MLD-048 (previously study rhASA-03 - NCT00633139) until HGT-1111 is commercially available or the study is terminated by the Sponsor, provided no safety concerns have emerged. The secondary objective of this study is to monitor disease progression and the safety profile of HGT-1111 administered to patients who have completed study HGT-MLD-048 (NCT00633139).

ELIGIBILITY:
Inclusion Criteria:

1. Subject's legally authorized guardian(s) must provide signed, informed consent prior to performing any study-related activities (Trial-related activities are any procedures that would not have been performed during normal management of the subject)
2. Completion of study HGT-MLD-048 (NCT00633139)
3. The subject and his/her guardian(s) must have the ability to comply with the protocol

Exclusion Criteria:

1. Spasticity so severe to inhibit transportation
2. Presence of known clinically significant cardiovascular, hepatic, pulmonary or renal disease or other medical condition that, in the opinion of the Investigator, would preclude participation in the trial
3. Any other medical condition or serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the trial

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2008-02-20 (Actual); Primary Completion 2010-10-22 (Actual); Study Completion 2010-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] I Dali C, Groeschel S, Moldovan M, Farah MH, Krageloh-Mann I, Wasilewski M, Li J, Barton N, Krarup C. Intravenous arylsulfatase A in metachromatic leukodystrophy: a phase 1/2 study. Ann Clin Transl Neurol. 2021 Jan;8(1):66-80. doi: 10.1002/acn3.51254. Epub 2020 Dec 17. PMID 33332761

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children with an established diagnosis of late metachromatic leukodystrophy (MLD) due to arylsulfatase A (ASA) deficiency were recruited.
Pre-assignment Details: All participants who completed Study HGT-MLD-048 (NCT00633139) participated in this study.
Groups:
- 100 U/kg HGT-1111: Participants received 100 units per kilogram (U/kg) of HGT1111 intravenous (IV) infusion every other week.
- 200 U/kg HGT-1111: Participants received 200 U/kg of HGT1111 IV infusion every other week.
Period: Overall Study
Arm/Group | 100 U/kg HGT-1111 | 200 U/kg HGT-1111
Started | 6 | 5
Completed | 3 | 1
Not Completed | 3 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 100 U/kg HGT1111: Participants received 100 U/kg of HGT1111 IV infusion every other week.
- 200 U/kg: Participants received 200 U/kg of HGT1111 IV infusion every other week.
- Total: Total of all reporting groups
Arm/Group | 100 U/kg HGT1111 | 200 U/kg | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 5 | 11
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] — Age at Week 54 or Week 56 in HGT-MLD-049 (NCT00681811)
  months | 53.14 (10.526) | 49.99 (8.752) | 51.71 (9.420)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 6 | 5 | 11

OUTCOME MEASURES:

1. Secondary Outcome: Level of Cerebrospinal Fluid (CSF) Sulfatide
Description: Level of CSF sulfatide measured at 6-month intervals in HGT-MLD-049 (NCT00681811).
Time Frame: Baseline until end of study (Week 139)
Population: Safety population. "Number of participants analysed" signifies participants who were evaluable for the respective arms under this outcome measure.
Measure: Mean (Standard Deviation); unit: nanomole per liter (nmol/L)
Groups:
- 100 U/kg HGT-1111 (Month 6): Participants received 100 U/kg of HGT1111 IV infusion every other week up to Month 6.
- 200 U/kg HGT-1111 (Month 6): Participants received 200 U/kg of HGT1111 IV infusion every other week up to Month 6.
- 100 U/kg HGT-1111 (Month 12): Participants received 100 U/kg of HGT1111 IV infusion every other week up to Month 12.
- 200 U/kg HGT-1111 (Month 12): Participants received 200 U/kg of HGT1111 IV infusion every other week up to Month 12.
- 100 U/kg HGT-1111 (Month 18): Participants received 100 U/kg of HGT1111 IV infusion every other week up to Month 18.
- 200 U/kg HGT-1111 (Month 18): Participants received 200 U/kg of HGT1111 IV infusion every other week up to Month 18.
- 100 U/kg HGT-1111 (Month 24): Participants received 100 U/kg of HGT1111 IV infusion every other week up to Month 24.
- 200 U/kg HGT-1111 (Month 24): Participants received 200 U/kg of HGT1111 IV infusion every other week up to Month 24.
Arm/Group | 100 U/kg HGT-1111 (Month 6) | 200 U/kg HGT-1111 (Month 6) | 100 U/kg HGT-1111 (Month 12) | 200 U/kg HGT-1111 (Month 12) | 100 U/kg HGT-1111 (Month 18) | 200 U/kg HGT-1111 (Month 18) | 100 U/kg HGT-1111 (Month 24) | 200 U/kg HGT-1111 (Month 24)
Number analyzed (Participants) | 5 | 4 | 5 | 3 | 3 | 3 | 1 | 2
nanomole per liter (nmol/L) | 685.0 (522.79) | 732.5 (545.06) | 745.0 (525.12) | 1150.0 (676.39) | 700.0 (526.78) | 850.0 (491.81) | 900.0 (NA) — Standard deviation could not be reported as there was only 1 evaluable participant. | 837.5 (441.94)

2. Secondary Outcome: Level of White Matter Metabolites
Description: Level of white matter metabolites [N-acetyl Aspartate (NAA)] measured at 6-month intervals in HGT-MLD-049 (NCT00681811).
Time Frame: Baseline until end of study (Week 139)
Population: Safety population. "Number of participants analysed" signifies participants who were evaluable for the respective arms under this outcome measure. No participants were analysed after Month 18, hence, data were not available after Month 18.
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- 200 U/Kg-HGT-1111(Month 6): Participants received 200 U/kg of HGT1111 IV infusion every other week up to Month 6.
- 100 U/kg- HGT-1111 (Month 12): Participants received 100 U/kg of HGT1111 IV infusion every other week up to Month 12.
- 100 U/kg- HGT-1111(Month 18): Participants received 100 U/kg of HGT1111 IV infusion every other week up to Month 18.
Arm/Group | 100 U/kg HGT-1111 (Month 6) | 200 U/Kg-HGT-1111(Month 6) | 100 U/kg- HGT-1111 (Month 12) | 200 U/kg HGT-1111 (Month 12) | 100 U/kg- HGT-1111(Month 18) | 200 U/kg HGT-1111 (Month 18)
Number analyzed (Participants) | 4 | 4 | 5 | 2 | 2 | 2
nmol/L | 0.528 (0.176) | 0.385 (0.237) | 0.598 (0.208) | 0.470 (0.198) | 0.510 (0.141) | 0.805 (0.445)

3. Secondary Outcome: Score of Gross Motor Function Measurement (GMFM)
Description: Gross motor function was measured using GMFM-88 at 6-month intervals. The GMFM-88 item scores were summed to calculate a total GMFM-88 score. For each GMFM-88 item, the score was between 0 (minimal) to 3 (maximum). The total GMFM-88 score was between 0 (minimal) to 264 (maximum). Decrease in GMFM score indicates disease progression.
Time Frame: Baseline until end of study (Week 139)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 100 U/kg HGT-1111 (Month 6) | 200 U/kg HGT-1111 (Month 6) | 100 U/kg HGT-1111 (Month 12) | 200 U/kg HGT-1111 (Month 12) | 100 U/kg HGT-1111 (Month 18) | 200 U/kg HGT-1111 (Month 18) | 100 U/kg HGT-1111 (Month 24) | 200 U/kg HGT-1111 (Month 24)
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 4 | 2 | 2 | 2
scores on a scale | 16.8 (11.30) | 9.2 (11.71) | 15.6 (15.84) | 8.7 (9.29) | 16.8 (13.60) | 9.0 (5.66) | 14.5 (10.61) | 13.0 (11.31)

4. Primary Outcome: Days of Exposure to HGT-1111
Description: End of study was defined as until HGT-1111 was commercially available, the participant's participation was discontinued, or the study was terminated by the Sponsor.
Time Frame: Baseline until end of study (Week 139)
Population: Safety population was defined as all enrolled participants who received at least one study infusion (or any portion of a dose) of HGT-1111.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- 100 U/kg HGT-1111: Participants received 100 U/kg of HGT1111 IV infusion every other week.
Arm/Group | 100 U/kg HGT-1111 | 200 U/kg HGT-1111
Number analyzed (Participants) | 6 | 5
Days | 644.7 (276.11) | 544.8 (397.27)

ADVERSE EVENTS:
Time Frame: Up to end of study (Week 139) which was defined as until HGT-1111 was commercially available, the patient's participation was discontinued, or the study was terminated by the Sponsor.
Description: All other adverse events (>5% reporting frequency) reported here are related to drug administration, all were infusion-related reactions.
Groups:
- 200 U/kg HGT1111: Participants received 200 U/kg of HGT1111 IV infusion every other week.
Arm/Group | 100 U/kg HGT1111 | 200 U/kg HGT1111
Serious Adverse Events (participants affected / at risk) | 2/6 | 4/5
Other Adverse Events (participants affected / at risk) | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 U/kg HGT1111 (N=6) | 200 U/kg HGT1111 (N=5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lower respiratory track infection (Infections and infestations) | 1 (3) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Catheter bacteraemia (Infections and infestations) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchitis acute (Infections and infestations) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 2 (3)
Pneumonia (Infections and infestations) | 0 (0) | 2 (3)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 U/kg HGT1111 (N=6) | 200 U/kg HGT1111 (N=5)
Pallor (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 3 (8)
Disease progression (General disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (16) | 4 (4)
Sleep disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1)
Phimosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Feeding tube complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood iron increased (Investigations) | 1 (1) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 1 (1) | 1 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (3)
Epilepsy (Nervous system disorders) | 1 (1) | 2 (3)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0)
Muscle spasticity (Nervous system disorders) | 2 (5) | 2 (3)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Conjunctival oedema (Eye disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (15) | 3 (10)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (9) | 3 (3)
Regurgitation of food (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urticaria generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (9) | 3 (6)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (13) | 2 (11)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (2)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis acute (Infections and infestations) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 3 (4) | 3 (4)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 2 (3)
Influenza (Infections and infestations) | 1 (2) | 1 (2)
Laryngitis (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (12) | 1 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (5) | 2 (4)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 1 (1)
Scarlet fever (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination due to lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days